CLINICAL TRIAL: NCT01234415
Title: Multicentric Pilot, Clinical Study of a Bone Substitute Safety and Efficacy in the Multi Traumatized Nasal Septum Reconstruction
Brief Title: Bone Substitute in the Multi Traumatized Nasal Septum Reconstruction
Acronym: NASEPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2010/16
Record Dates: First submitted 2010-11-02; First posted 2010-11-04 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Nasal Septum
Keywords: nasal; septum; reconstruction
MeSH Terms: interventions — Rhinoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patient (Experimental)
  Interventions: Device: Rhinoplasty

INTERVENTIONS:
Device: Rhinoplasty — Rhinoplasty is performed under general anaesthesia; the duration is 1 to 2 hours. The surgical approach for implantation of the biomaterial is external rhinoplasty. The incision is made at the columella (base of nose) and becomes internal for the scar to be as unobtrusive as possible. The septum skeleton is then destroyed in order to place the synthetic biomaterial. The biomaterial is remodelled in order to have a natural external aspect of the nose. The incision is closed and the wicks are put in place in the nose for 4 days. A cast and a sticker will be put in place after surgery to maintain properly the biomaterial.

SUMMARY:
The aim of this project is to evaluate the safety and efficacy of the biomaterial made of HAP/TCP (BCP, Kasios®), in septoplasties of multi traumatized human nose. The use of this biomaterial will avoid the graft sampling and we expect it to be a good substitute to support the nasal pyramid while favouring the respiratory epithelium regeneration. Thus, that would confirm previous in vitro and in vivo studies.

DETAILED DESCRIPTION:
Five to ten percent of the post-traumatic septo-rhinoplasties require a total reconstruction of the septal skeleton. This surgery requires using autologous bone graft (iliac, costal, or parietal). However these swabs include surgical risks, have a particular morbidity non negligible and particular quality imperfections (resorption level, texture, shape, integration) requiring a complex and long lasting shaping before implantation. To avoid the using of bone graft, a large scale of products has been developed to propose a synthetic bone substitute as a support for bone reconstruction. The bone substitute, BCP, made of hydroxyl apatite (HAP) and tricalcium phosphate (TCP), is thus largely used in orthopaedics, and CE marked in numerous indications (like sinus lift). The stake is to validate that it can be used in septo-rhino-plasties. This septic zone presents characteristics which required in vitro and in vivo studies, showing that the conclusions are a good biocompatibility of BCP for human epithelial cells and in septal area of rabbits and sheep. The ultimate step to validate this concept consists in conducting a pilot clinical study on 25 patients with the indication of septoplasties to verify its safety and efficacy in clinical conditions. This study will have an 18 months inclusion period and 6 months of follow up. The principal objective is to assess the HAP/TCP biomaterial safety and to confirm clinically and histologically the good affinity of human epithelial cells for this material. Secondary objective is to demonstrate that the restoration of the normal nasal anatomy with the material re-establishes the nasal respiratory shape and function. Clinical data, questionnaires, and photos will be collected pre operatively and at day 4, 10, and month 2 and 6 after surgery. The endonasal biopsy and fiberoptic endoscopy will be realised at 2 and 6 months post operatively and will be supplementary to the routine care protocol of the surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 60
* Indication of tissue replacement in a nasal septum, which skeleton is lacking or non usable for patients having:
* Paradoxal nasal obstruction with saddle nose type III and IV or flabby nose
* Nasal obstruction with an obstacle caused by a moved multifracture skeleton
* Written informed consent
* Patient with social insurance

Exclusion Criteria:

* Post-menopausal women : lack of efficient contraception (intra uterine dispositive or contraceptive pill)
* Breast feeding or pregnant women
* HIV or VHB or VHC seropositive subject
* Inflammatory or infectious active rhino sinusitis
* Nasal an sinus surgery or trauma ended from less than 8 months
* Toxic medicated Rhinitis to vasoconstrictors
* Diabetic : all type of diabetes (without or with therapy)
* Non treated cardiac disease
* Any contra indication to surgery
* Any contra indication to the biomaterial use like evolutive infection, bone disease or local necrosis
* Radiotherapy antecedent of the cephalic and cervical extremity
* Local or regional therapy with corticoids currently, or stopped from less than 2 months
* Patient participating to another study with an exclusion period still going on during pre-inclusion period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Safety | up to 6 months after surgery
  Frequency and severity of expected Adverse and Severe Adverse Events, as material extrusion, infection (wall abscess), and chronic pathological inflammatory reaction, pain, epistaxis.
Epithelial cells affinity | up to 6 months after surgery
  macroscopic mucous membrane integrity (ciliated cells), absence of perforation, pathological analyses of biopsy to research sub epithelial infiltration, respiratory epithelial differentiation markers (HES, MOVAT pentachrome), immunohistochemistry (AB against cytokeratines 7, 8, 19, UEA1, MUC5AC) and MEB, MET analyses.

SECONDARY OUTCOMES:
Performance with Internal and external nasal shape assessment | month 2 and 6 after surgery.
  Photography and fiberoptic endoscopy
Performance with Functional Performance Assessment | pre operatively and post operatively at day 4, 10, and month 2 and 6 after surgery.
  NOSE and RHINO quality of life questionnaires Clinical data, questionnaires, and photos will be collected pre operatively and post operatively at day 4, 10, and month 2 and 6 after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic LE TAILLANDIER de GABORY, Dr, Principal Investigator — University Hospital, Bordeaux
Locations (3):
- France (3):
  - Service d'Oto-rhino-laryngologie et Chirurgie cervico-faciale - CHU de Bordeaux, Bordeaux
  - Service d'Oto-rhino-laryngologie - Clinique St Augustin, Bordeaux
  - Service d'Oto-rhino-laryngologie - Hôpital Dupuytren, Limoges